CLINICAL TRIAL: NCT07054606
Title: A Phase 4, Multicenter, Open-Label Study to Evaluate Concomitant Perfluorohexyloctane Use With Contact Lens Wear
Brief Title: A Study to Evaluate Concomitant Perfluorohexyloctane Use With Contact Lens Wear
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BL-RX01-BAJA-1403
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Miebo (perfluorohexyloctane ophthalmic solution) (Experimental)
  Interventions: Drug: Perfluorohexyloctane ophthalmic solution

INTERVENTIONS:
Drug: Perfluorohexyloctane ophthalmic solution — Eligible subjects will receive Miebo up to 4 times bilaterally on Day 1/Visit 1 (1 drop instilled bilaterally by site staff in-clinic while wearing contact lenses and the rest self-administered throughout the remainder of the day while wearing contact lenses). Starting on Day 2, subjects will self-administer the first drop of Miebo bilaterally before inserting contact lenses for the day. Subjects will wait 30 minutes after the first dose of Miebo to insert their contact lenses and will then instill 3 additional drops of Miebo while wearing contact lenses approximately evenly spaced throughout the rest of the day. Subjects will continue to self-administer Miebo QID bilaterally following the dosing schedule from Day 2 for approximately 30 days. Subjects are expected to record daily VAS assessments throughout the study. The VAS assessments will be collected by the sites at Visits 2, 3, and 4.

SUMMARY:
Assess the impact of concomitant Miebo use while wearing contact lenses

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of consent
2. Able to provide written voluntary informed consent and sign the Health Insurance Portability and Accountability Act (HIPAA) form as well as the Experimental Subjects Bill of Rights(for subjects in California)
3. Subject must have a documented Manifest Refraction by the PI (or sub-investigator at the same site) performed in the past 180 days prior to screening.
4. Currently wearing soft, frequent-replacement lenses bilaterally (daily-disposable, bi-weekly, or monthly lenses that are available in the US), that have been worn habitually for a minimum of 5 days/week for 6 hours/day over the last 6 months prior to Visit 1 and is willing to wear them for at least 6 hours/day every day during the study (i.e., 30 consecutive days of contact lens wear). Almost all soft contact lenses qualify for study (see exclusion criterion #2 below).
5. Achieves acceptable lens fit as well as ETDRS VA correctable with contact lenses to +0.20 logMAR or better in each eye at Visit 1
6. Able and willing to follow instructions, including participation in all trial assessments and visits
7. Be willing to submit to urine pregnancy test at Visits 1 and 4 for female subjects of childbearing potential.
8. Female subjects of childbearing potential must agree to use 1 medically acceptable method of birth control; acceptable methods of contraception include hormonal (oral, implantable, injectable, or transdermal) contraception; mechanical (spermicide in conjunction with a barrier such as a diaphragm or condom) contraception; intrauterine device; or surgical sterilization of partner. True abstinence may be regarded as an acceptable method of birth control (when this is in line with the preferred and usual lifestyle of the subject); however, if the subject becomes sexually active during the trial, she must use an acceptable method of birth control as defined above for the remainder of the trial. Note: Females of childbearing potential include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy).
9. Male subjects with a female partner of childbearing potential, must use at least 1 medically acceptable method of birth control. Note: Acceptable methods of birth control are true abstinence (when this is in line with the preferred and usual lifestyle of the subject) or vasectomy at least 3 months prior to receiving Investigational Product. Without a vasectomy, condoms with spermicide must be used throughout the study duration.

Exclusion Criteria:

1. Subjects who do not have a documented Manifest Refraction within 180 days prior to Visit 1 by the Principal Investigator (or sub-investigator at the same site).
2. Subjects who are non-contact lens wearers or who have changed contact lens type/brand within the last 6 months
3. Subjects who wear scleral lenses, rigid gas-permeable lenses, hybrid lenses, custom soft contact lenses with a replacement schedule >30 days, or soft contact lenses on an extended-wear basis (i.e., AirOptix Night and Day contact lenses and other lenses approved for overnight wear)
4. Have any clinically significant ocular surface slit-lamp findings in either eye and/or, in the opinion of the Investigator, have any findings that could interfere with trial parameters or impact a subject's ability to wear contact lenses throughout the study, including:

   1. History of Stevens-Johnson syndrome
   2. Active blepharitis or lid margin inflammation
   3. Dry eye disease secondary to scarring, irradiation, alkali burns, cicatricial pemphigoid, or destruction of conjunctival goblet cells (as with vitamin A deficiency)
   4. Abnormal lid anatomy causing incomplete eyelid closure
   5. Abnormal cornea shape (keratoconus)
   6. Corneal epithelial defect or significant confluent staining or filaments
   7. History of ocular malignancy
5. Pterygium or pinguecula in either eye that, in the opinion of the Investigator, could interfere with fit of a soft contact lens
6. Use of any of the following ocular therapies in either eye within 30 days prior to Visit 1: Vuity®, topical ocular steroid treatments, topical antibiotics, topical anti-allergy medications, prescription dry eye therapy including varenicline nasal spray, or topical anti-glaucoma medication
7. Use of any eye drops (prescription or over-the-counter, such as artificial tears, re-wetting drops, RYZUMVITM, or Lumify®) and/or TrueTear™ device (intranasal tear neurostimulator) in either eye within 24 hours prior to Visit 1, or plan to use these therapies during the course of the study
8. Have active uncontrolled ocular allergies or ocular allergies that are expected to be active during the trial period
9. Have undergone intraocular surgery or ocular laser surgery in either eye within 3 months prior to Visit 1; have undergone refractive surgery in either eye within 1 year prior to Visit 1
10. Planning to undergo an ocular surgical intervention (e.g., intraocular surgery, ocular surgery, cataract surgery, LASIK, etc.) in either eye during the trial period.
11. Have active ocular or systemic infection (bacterial, viral, or fungal), including fever
12. Be unwilling to submit to a urine pregnancy test at Visits 1 and 4 for women of childbearing potential. Note: Females of childbearing potential include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy).
13. Female subjects who are pregnant, nursing, or planning a pregnancy
14. Female subjects of childbearing potential who are not using 1 acceptable method of birth control; acceptable methods of contraception include hormonal (oral, implantable, injectable, or transdermal) contraception; mechanical (spermicide in conjunction with a barrier such as a diaphragm or condom) contraception; intrauterine device; or surgical sterilization of partner. True abstinence may be regarded as an acceptable method of birth control; however, if the subject becomes sexually active during the trial, she must agree to use 1 acceptable method of birth control as defined above for the remainder of the trial
15. Male subjects with a female partner of childbearing potential, who is not willing to use 1 acceptable method of birth control throughout the study. Note: Acceptable methods of birth control are true abstinence (when this is in line with the preferred and usual lifestyle of the subject) or unwilling to use condoms with spermicide if he has not had a vasectomy at least 3 months prior to receiving Investigational Product.
16. Have an uncontrolled systemic disease that, in the opinion of the Investigator, will interfere with the trial
17. Have a known allergy and/or sensitivity to the Investigational Product or diagnostic substances (e.g., fluorescein) to be used in the study
18. Are currently enrolled in any investigational drug or device study or have used Miebo within 30 days prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline (CFB) in CLDEQ-8 score at Visit 4 | Assessed for approximately 30 days
  Unabbreviated scale title: Contact Lens Dry Eye Questionnaire-8 Min: 1 Max: 37 Higher scores mean worse.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Site 101, San Diego, California
  - Site 107, Longwood, Florida
  - Site 104, Pittsburg, Kansas
  - Site 102, Medina, Minnesota
  - Site 108, Vestal, New York
  - Site 103, Athens, Ohio